CLINICAL TRIAL: NCT00000194
Title: Neurobiology of Opioid Dependence: 3
Brief Title: Neurobiology of Opioid Dependence: 3 - 3
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-00191-3; K20DA000191 (NIH); K20-00191-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2015-08

CONDITIONS: Opioid-Related Disorders
Keywords: opioid disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Cycloserine

INTERVENTIONS:
Drug: Cycloserine

SUMMARY:
The purpose of this study is to study the effects of cycloserine on naloxone-precipitated opiate withdrawal.

ELIGIBILITY:
Please contact site for information.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1993-01; Primary Completion 1998-01 (Actual); Study Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
Behavioral, subjective, measures of naloxone-preci
Phsyiological, neuroendocrine measures of naloxone

CONTACTS AND LOCATIONS:
Overall Officials: Marc I Rosen, M.D., Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, New Haven, Connecticut, United States